CLINICAL TRIAL: NCT02507544
Title: A Phase I Safety and Pharmacokinetic Study of TRX-818 Administered Orally to Patients With Advanced Cancer
Brief Title: A Safety and Pharmacokinetic Study of TRX-818 Administered Orally to Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TaiRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVM-001
Record Dates: First submitted 2015-07-15; First posted 2015-07-24 (Estimated); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Carcinoma; Advanced Cancer
Keywords: Advanced Solid Malignancy; Safety and Tolerability; Tumor Response; Hematology; Oncology
MeSH Terms: conditions — Carcinoma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TRX-818 (Experimental)
  Interventions: Drug: TRX-818 capsules

INTERVENTIONS:
Drug: TRX-818 capsules

SUMMARY:
TRX-818 is a new small molecule chemical entity being developed as a potential anti-cancer therapeutic by TaiRx, Inc. TRX-818 is a potent anti-cancer agent in numerous human cancer cell lines. The objectives of this study are to determine the safety profile of TRX-818 including identification of dose limiting toxicity (DLT) and maximum tolerated dose (MTD) and determine the recommended dose and regimen(s) to initiate Phase 2.

ELIGIBILITY:
Inclusion Criteria:

1. Tumor eligibility:

   Histologically confirmed advanced malignancies refractory to standard of care therapy, or for whom no standard of care therapy is available.
2. Solid tumors must have measurable or evaluable disease as per Response Evaluation Criteria in Solid Tumors (RECIST v. 1.1). Target lesions that have been previously irradiated will not be considered measurable (lesion) unless increase in size is observed following completion of radiation therapy. Leukemia, lymphomas and multiple myeloma must have measurable disease as per response criteria.
3. Female or male, 18 years of age or older.
4. Eastern Cooperative Oncology Group performance status 0 to 2. Resolution of all acute toxic effects of prior therapy or surgical procedures to grade 1 (except alopecia).
5. Adequate organ function as defined by the following criteria:

   * Serum aspartate transaminase (AST) and serum alanine transaminase (ALT) ≤3 x upper limit of normal (ULN), or AST and ALT ≤5 x ULN if liver function abnormalities are due to underlying malignancy
   * Total serum bilirubin ≤1.5 x ULN (except for patients with documented Gilbert's syndrome)
   * Absolute neutrophil count (ANC) >= 1500/µL
   * Platelets >= 90,000/µL
   * Hemoglobin >= 9.0 g/dL
   * Serum creatinine ≤2.0 x ULN
6. Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all the pertinent aspects of the trial prior to enrollment.
7. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

Patients presenting with any of the following will not be included in the trial:

1. Major surgery, radiation therapy, or systemic anti-cancer therapy within 4 weeks of starting study treatment.
2. Prior high-dose chemotherapy requiring hematopoietic stem cell rescue except for patients with lymphoma or myeloma.
3. Current treatment on another clinical trial.
4. Brain metastases, spinal cord compression, carcinomatous meningitis, or leptomeningeal disease unless appropriately treated and neurologically stable for at least 4 weeks.
5. Any of the following within the 12 months prior to starting study treatment: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, congestive heart failure, or cerebrovascular accident including transient ischemic attack; within 6 months prior to starting study treatment for pulmonary embolus. However, upon agreement between the investigator and sponsor, the 6 month post-event-free period for a patient with a pulmonary embolus can be waived if due to advanced cancer. Appropriate treatment with anticoagulants is permitted.
6. Hypertension that cannot be controlled by medications (>150/100 mmHg despite optimal medical therapy).
7. Current treatment with therapeutic doses of warfarin (low dose warfarin up to 2 mg Per oral (PO) daily for deep vein thrombosis prophylaxis is allowed).
8. Known human immunodeficiency virus infection.
9. Pregnancy or breastfeeding. Female patients must be surgically sterile or be postmenopausal, or must agree to the use of effective contraception during the period of therapy. All female patients with reproductive potential must have a negative pregnancy test (serum or urine) prior to enrollment. Male patients must be surgically sterile or must agree to use effective contraception during the period of therapy. The definition of effective contraception will be based on the judgment of the principal investigator or a designated associate.
10. Other severe acute or chronic medical or psychiatric conditions or laboratory abnormalities that would impart, in the judgment of the investigator and/or sponsor, excess risk associated with study participation or study drug administration, which would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-04-29 (Actual); Study Completion 2019-05-20 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) of TRX-818 | up to 28 days
  Toxicities will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.0.
Maximum tolerated dose (MTD) of TRX-818 | up to 28 days
  The MTD will be defined as the dose level at which at most one of six patients experiences a DLT after 28 days of treatment have occurred, with the next higher dose having at least 2/3 or 2/6 patients experiencing a DLT.

SECONDARY OUTCOMES:
Preliminary assessment of anti-tumor activity by Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST 1.1) | up to 112 days
Composite measure of pharmacokinetics (PK) parameters of TRX-818 and its metabolites TRX-818M1 to include AUC(0-last), Cmax, Tmax, T(1/2). | Selected time points during first 28 days
  AUC(0-last): area under the plasma concentration versus time curve to the time of the last measurable concentration; Cmax: maximum plasma concentration; Tmax: time to maximum plasma concentration; T(1/2): terminal elimination half-life
Time to tumor progression (TTP) | up to 112 days

CONTACTS AND LOCATIONS:
Overall Officials: Anthony W Tolcher, M.D., FRCP(C), Principal Investigator — South Texas Accelerated Research Therapeutics, LLC (START); Nehal Lakhani, M.D., Ph.D., Principal Investigator — START Midwest
Locations (2):
- United States (2):
  - START Midwest, Grand Rapids, Michigan
  - South Texas Accelerated Research Therapeutics, LLC (START), San Antonio, Texas